CLINICAL TRIAL: NCT01544686
Title: Chlorhexidine Containing Iv-securement Dressings for the Prevention of Central Venous Catheter-related Blood Stream Infections in Neutropenic Patients: a Randomized Trial
Brief Title: Antimicrobial Catheter Securement Dressings for the Prevention of Cvc-related Bloodstream Infections in Cancer Patients
Acronym: COAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, Principal Investigator, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DRKS00003368
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Bloodstream Infection
Keywords: neutropenia; cancer; fever; central venous catheter; infection
MeSH Terms: conditions — Sepsis; Neutropenia; Neoplasms; Fever; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3M™ Tegaderm CHG IV (Active Comparator): Patients receive the 3M Tegaderm CHG IV securement dressing after placement of a central venous catheter.
  Interventions: Device: 3M™ Tegaderm™ CHG IV and 3M™ Tegaderm™ Advanced IV
- 3M™ Tegaderm™ Advanced IV' (Placebo Comparator): Patients receive the 3M Tegaderm Advanced IV securement dressing after placement of a central venous catheter.
  Interventions: Device: 3M™ Tegaderm™ CHG IV and 3M™ Tegaderm™ Advanced IV

INTERVENTIONS:
Device: 3M™ Tegaderm™ CHG IV and 3M™ Tegaderm™ Advanced IV — Patients receive the 3M™ Tegaderm CHG IV securement dressing or the 3M Tegaderm Advanced IV securement dressing after placement of a central venous catheter.

SUMMARY:
In neutropenic cancer patients, catheter-related bloodstream infections may cause severe infections and even death. To assess the prophylactic effect of a chlorhexidine coated catheter securement dressing on the incidence of catheter-related bloodstream infections, this open, randomized trial is being carried out. CHG iv Tegaderm securement dressing will be randomized in a 1:1 fashion against Tegaderm Advanced iv securement dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a central venous catheter for chemotherapy of AML or ALL
* Patients receiving a central venous catheter for high-dose chemotherapy with consecutive autologous stem cell transplantation or any other condition with an expected duration of chemotherapy-associated neutropenia of at least 5 days and an expected duration of central venous catheter use of at least 10 days
* Age >= 18 years

Exclusion Criteria:

* Condition with an expected duration of chemotherapy-associated neutropenia of at less than 5 days and an expected duration of central venous catheter use of less than 10 days
* Use of a central venous catheter with antimicrobial coating other than chlorhexidine and/or silver-sulfadiazine
* Limited venous status, impeding acquisition of peripheral blood cultures in case of febrile neutropenia
* Patients previously enrolled in the study
* Tunneled central venous catheters
* Shaldon catheters
* CVC insertion via the V. femoralis
* Fever (T > 37.8°C) related to a suspected or confirmed bacterial infection at randomization
* Known allergic/hypersensitivity reaction to any compounds of the treatment
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of definite catheter-related bloodstream infection during the first 14 days after placement of the central venous catheter | 14 days
  Incidence of definite catheter-related bloodstream infection during the first 14 days after placement of the central venous catheter

SECONDARY OUTCOMES:
Incidence of definite catheter related bloodstream infection-related severe sepsis during the first 14 days after placement of the central venous catheter | 14 days
  Incidence of definite catheter related bloodstream infection-related severe sepsis during the first 14 days after placement of the central venous catheter
Definite catheter-related bloodstream infection-related mortality during the first 14 days after placement of the central venous catheter | 14 days
  Definite catheter-related bloodstream infection-related mortality during the first 14 days after placement of the central venous catheter
Overall incidence of catheter-related bloodstream infection | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Overall incidence of catheter-related bloodstream infection (evaluated by definite, probable and proven criteria)
Overall catheter-related bloodstream infection-related severe sepsis | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Overall catheter-related bloodstream infection-related severe sepsis (evaluated by definite, probable and proven criteria)
Overall catheter-related bloodstream infection-related mortality | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Overall catheter-related bloodstream infection-related mortality(evaluated by definite, probable and proven criteria)
Overall mortality | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Overall mortality
Time to removal of central venous catheter | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Time to removal of central venous catheter
Time to central venous catheter-related blood stream infections | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Time to central venous catheter-related blood stream infections
Time to first neutropenic fever | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Time to first neutropenic fever
Rate of unplanned changes | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Rate of unplanned changes of the catheter securement dressing.
Tolerability/safety | From placement of the central venous catheter until the follow-up at a maximum of 56 days
  Tolerability/safety is defined as the number of toxicity-related study therapy discontinuations.

CONTACTS AND LOCATIONS:
Overall Officials: Maria JG Vehreschild, Dr. med., Principal Investigator — University Hospital of Cologne
Locations (5):
- Germany (5):
  - Klinikum Schwabing, Munich, Bavaria
  - Klinikum Neuperlach, Munich, Bavaria
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Universitätsmedizin Berlin - Charité, Berlin, State of Berlin

REFERENCES:
- [Derived] Schalk E, Teschner D, Hentrich M, Boll B, Panse J, Schmidt-Hieber M, Vehreschild MJGT, Biehl LM. Central venous catheter-related bloodstream infections in patients with hematological malignancies: Comparison of data from a clinical registry and a randomized controlled trial. Infect Control Hosp Epidemiol. 2020 Feb;41(2):254-256. doi: 10.1017/ice.2019.335. No abstract available. PMID 31818338
- [Derived] Schalk E, Biehl LM, Farber J, Schluter D, Vehreschild MJGT, Fischer T. Determination of a Cutoff Time Point for Prophylactic Exchange of Central Venous Catheters for Prevention of Central Venous Catheter-Related Bloodstream Infections in Patients with Hematological Malignancies. Infect Control Hosp Epidemiol. 2017 Jul;38(7):888-889. doi: 10.1017/ice.2017.92. Epub 2017 May 18. No abstract available. PMID 28514979
- [Derived] Biehl LM, Huth A, Panse J, Kramer C, Hentrich M, Engelhardt M, Schafer-Eckart K, Kofla G, Kiehl M, Wendtner CM, Karthaus M, Ullmann AJ, Hellmich M, Christ H, Vehreschild MJ. A randomized trial on chlorhexidine dressings for the prevention of catheter-related bloodstream infections in neutropenic patients. Ann Oncol. 2016 Oct;27(10):1916-22. doi: 10.1093/annonc/mdw275. Epub 2016 Jul 25. PMID 27456299